CLINICAL TRIAL: NCT06152939
Title: Relation of Laboratory Indices to Left Ventricular Thrombus Formation in Patients With Acute Anterior ST Segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention or Thrombolytic Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Al zahraa Sayed Mahmoud Mohamed, Relation of laboratory indices to left ventricular thrombus formation in patients with acute anterior ST segment elevation myocardial infarction undergoing primary percutaneous coronary intervention or thrombolytic therapy, Assiut University
Other Study IDs: LV thrombus in anterior STEMI
Record Dates: First submitted 2023-09-19; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Left Ventricular Thrombus
MeSH Terms: interventions — Thrombolytic Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: patients with acute anterior ST segment elevation myocardial infarction undergoing primary percutaneous coronary intervention .
  Interventions: Other: Primary percutaneous coronary intervention or thrombolytic therapy
- 2: patients with acute anterior ST segment elevation myocardial infarction have thrombolytic therapy .
  Interventions: Other: Primary percutaneous coronary intervention or thrombolytic therapy

INTERVENTIONS:
Other: Primary percutaneous coronary intervention or thrombolytic therapy — Primary percutaneous coronary intervention or thrombolytic therapy

SUMMARY:
• to find the relationship between the different hematological indices including platelet indices, and blood cell ratios, to the development of LV thrombus in acute anterior STEMI patients managed by primary percutaneous coronary intervention (PPCI) , or thrombolytic therapy .

DETAILED DESCRIPTION:
ST-segment elevation myocardial infarction (STEMI) has been associated with a high rate of morbidity and mortality (1) Left ventricular thrombus (LVT), one of the most common complications of acute anterior myocardial infarction is linked to the potentially devastating outcome of thromboembolism or stroke [1, 2] , In the era of primary PCI, despite aggressive reperfusion treatment and antithrombotic treatment, the presence of LVT remains high after anterior STEMI), Determining the correlation between clinical and laboratory indicators of thrombosis is the key to the prevention of thromboembolism , The PLR( platelets to lymphocytes ratio ), a new index , provides information about both the inflammatory and thrombosis pathways(3), It is known since long that larger platelets are metabolically and enzymatically more active than small platelets and they have higher thrombotic potentials , that is why MPV , Platelets count , and platelet crit (PCT) are related to platelets activation and they have been suggested as markers of haemostasis , Increase MPV is thought to be associated with thrombus formation in all vascular structures , Recent evidence has shown the meaningful clinical information of the PLR in coronary heart disease and thrombotic diseases (whether diagnostic information or prognostic information). Despite the findings above, data regarding the role of this inflammatory biomarker in LVT are lacking. We conducte a prospective case-control study to explore the correlation between LVT and the PLR and different hematologic indices among anterior STEMI patients with LV dysfunction after primary PCI, or thromolytic therapy, Hematological markers, predictive and even diagnostic value in cardiovascular diseases (CVDs) is a major field of research (4) Leukocytes are considered essential for thrombus formation as well as plaque activation in acute coronary syndrome (ACS). The most reliable indicator of unfavorable outcomes has been proven to be platelet count and may platelet volume, haematocrit, haemoglobin, peak level Troponin and CK-MB (5), Monocytes play a critical role in atherosclerosis by releasing cytokines that are pro-inflammatory and pro-oxidant (6) High values of the monocyte are associated with unfavourable outcomes and severe coronary artery disease (7) ). So, we aimed to find relationship between the different hematological indices and LV thrombus formation in anterior STEMI managed by primary percutaneous coronary intervention (PPCI) or thrombolytic therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients presented to Assiut university cardiac catheterization laboratory with acute anterior STEMI and managed with PPCI or thrombolytic therapy.

Exclusion Criteria:

* • Patients not eligible to PPCI

  * Patients presented with inferior or lateral STEMI or any type of STEMI other than anterior STEMI.

Ages: 15 Years to 95 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients present with acute anterior STEMI and undergoing primary percutaneous coronary intervention or thrombolytic therapy in Assiut university heart hospital (AUHH). Patients will be categorized into 2 groups: those with LVT and those without LVT development.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
the relation of different hematological indices to the development of LV thrombus in acute anterior STEMI patients managed by primary percutaneous coronary intervention (PPCI) or thrombolytic therapy . | baseline
  • To assess the relation of different hematological indices including platelet indices: Mean platelet volume (MPV), Mean platelet component (MPC) , Plateletcrit (PCT), platelet distribution width (PDW), Mean platelet mass (MPM), and blood cell ratios: Neutrophil to lymphocyte ratio (NLR), Platelet to lymphocyte ratio (PLR),White blood cell to Mean platelet volume (WMR) to the development of LV thrombus in acute anterior STEMI patients managed by primary percutaneous coronary intervention (PPCI) or thrombolytic therapy .

SECONDARY OUTCOMES:
o Assessment of protein C, S, and activated protein C resistance (APCR) and its relation to LVT development. | baseline
  * Assessment of protein C, S, and activated protein C resistance (APCR) and its relation to LVT development.
  * Relation of the former indices to intracoronary thrombus burden
  * Relation of the former indices to major adverse cardiac and cerebrovascular events (MACCEs), both in-hospital and at 3 months

REFERENCES:
- See also: Related Info — https://www.google.com/search?q=Chacon-Diaz+M%2C+Custodio&rlz=1C1RLNS_enEG1029EG1029&oq=Chacon-Diaz+M%2C+Custodio&aqs=chrome..69i57j33i10i160.56552j0j15&sourceid=chrome&ie=UTF-8
- See also: Related Info — https://www.google.com/search?q=vogel+b+claessen+e+arnold+v+et+al+2019%29&sca_esv=566650974&rlz=1C1RLNS_enEG1029EG1029&ei=NNwJZdGRNeKrkdUPq8uu4Ak&oq=Vogel+B%2C+Claessen+E%2C+Arnold+V+et+al+2019&gs_lp=Egxnd3Mtd2l6LXNlcnAiKFZvZ2VsIEIsIENsYWVzc2VuIEUsIEFybm9sZCBWIGV0IGFsIDIwMTkqAggAMgUQIRigAUisnAhQsPYBWL-UB3AFeACQAQGYAcYDoAGyO6oBCjAuMzYuNC4xLjG4AQHIAQD4AQGoAgDCAgsQABiABBixAxiDAcICERAuGIAEGLEDGIMBGMcBGNEDwgIIEAAYgAQYsQPCAgsQLhiKBRixAxiDAcICBRAAGIAEwgIOEC4YgAQYsQMYxwEY0QPCAg0QLhiKBRjHARjRAxhDwgIgEC4YgAQYsQMYgwEYxwEY0QMYlwUY3AQY3gQY4ATYAQHCAg0QABiKBRixAxiDARhDwgILEC4YgAQYxwEY0QPCAgUQLhiABMICCxAuGIAEGMcBGK8BwgIUEC4YgAQYlwUY3AQY3gQY3wTYAQHCAgYQABgWGB7CAgkQABgWGB4Y8QTCAggQIRgWGB4YHcICBxAhGKABGArCAgQQIRgVwgIFEAAYogTiAwQYACBBiAYBugYGCAEQARgU&sclient=gws-wiz-serp
- See also: Related Info — https://www.google.com/search?q=kumar+v+sharma+k+kumar+t+2020+pdf&sca_esv=566650974&rlz=1C1RLNS_enEG1029EG1029&ei=ct8JZfnjGP2ikdUPnOCb6Aw&oq=Kumar+V%2C+sharma+K+%2CKumar+T+2020&gs_lp=Egxnd3Mtd2l6LXNlcnAiH0t1bWFyIFYsIHNoYXJtYSBLICxLdW1hciBUIDIwMjAqAggAMgcQIRigARgKSK-6BVDADli-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_CAggQIRgWGB4YHcICChAhGBYYHhgPGB3CAgQQIRgV4gMEGAEgQYgGAboGBggBEAEYFA&sclient=gws-wiz-serp